CLINICAL TRIAL: NCT01127256
Title: Comparative Study of Zonisamide and Carbamazepine as an Initial Monotherapy: Efficacy and Safety Evaluation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Korea Inc. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2090-S082-405
Record Dates: First submitted 2010-05-19; First posted 2010-05-20 (Estimated); Results first posted 2012-07-26 (Estimated); Last update posted 2022-01-04 (Actual); Status verified 2010-05

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Zonisamide; Carbamazepine

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: zonisamide
- 2 (Active Comparator)
  Interventions: Drug: carbamazepine

INTERVENTIONS:
Drug: zonisamide — Initial dose was 100mg/day, increased by 100mg. The maximum dose was 600mg/day.
  Arms: 1
Drug: carbamazepine — Initial dose was 100mg/day, increased by 200mg every 1 week to 600mg/day. The maximum dose was 1200mg/day.
  Arms: 2

SUMMARY:
The purpose of this study is to compare the efficacy and safety of zonisamide with carbamazepine and to determine the optimum dose of zonisamide in patients with epilepsy.

DETAILED DESCRIPTION:
To compare efficacy and safety between the zonisamide group and the carbamazepine group. The zonisamide group will be divided into 2 subgroups: Slow-titration group and Fast-titration group to find out optimum titration of zonisamide. This study will proceed through 25~27 weeks.

ELIGIBILITY:
Inclusion criteria:

1. Epilepsy patients over 15 years old.
2. Occurrence of seizure should be more than one time within recent 3 months and more than two times within recent 6 months.
3. Patients who have not taken antiepileptic drugs (AEDs) in recent 3 months.
4. Female who can be in the month of pregnancy should agree to prevent conception.
5. Patients who agree with Informed Consent Form.

Exclusion criteria:

1. Patients who have Myoclonic seizures and/or Absence seizures.
2. Patients who have progressive central nervous system (CNS) disorder.
3. Patients who have serious systemic disorder.
4. Upward of doubled normal serum glutamic oxaloacetic transaminase (SGOT) or serum glutamic pyruvic transaminase (SGPT) level and/or tripled blood urea nitrogen (BUN)/Creatinine levels.
5. Patients who have renal stones.
6. Medical history of medicinal poisoning and/or alcoholism.
7. Patients who have long-term medication history (more than 6 months) of zonisamide and/or carbamazepine.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2006-05-31 (Actual); Primary Completion 2009-05-31 (Actual); Study Completion 2009-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jihee Mun, Study Director — Medical Department, Eisai Korea Inc.
Locations (12):
- South Korea (12):
  - Seoul National Univ. Bundang Hosp., Bundang
  - Dongguk Univ. Ilsan Hosp., Ilsan
  - Inha Univ. Hosp., Incheon
  - Chungnam National Univ. Hosp., Jungnam
  - Boramae Medical Center, Seoul
  - Eulji General Hosp., Seoul
  - Ewha Womans Univ. Mokdong Hospital, Seoul
  - Hallym Univ. Medical Center, Seoul
  - Hanyang Univ. Medical Center, Seoul
  - Konkuk Univ. Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National Univ. Hosp., Seoul

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was recruited at 12 centers in Korea during the period of May 2006 to May 2009.
Groups:
- Zonisamide: Initial dose was 100 mg/day, increased by 100 mg. The maximum dose was 600 mg/day.
Period: Overall Study
Arm/Group | Zonisamide | Carbamazepine
Started | 96 | 104
Completed | 57 | 65
Not Completed | 39 | 39
Not completed — Adverse Event | 13 | 13
Not completed — Lack of Efficacy | 4 | 0
Not completed — Lost to Follow-up | 16 | 17
Not completed — Withdrawal by Subject | 5 | 9
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zonisamide | Carbamazepine | Total
Number analyzed (Participants) | 96 | 104 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (15.9) | 35.7 (15.1) | 37.7 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 53 | 102
  Male | 47 | 51 | 98
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 96 | 104 | 200
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants With Seizure Free Rate
Description: The percentage of participants who had no seizure during the trial.
Time Frame: 24 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Zonisamide | Carbamazepine
Number analyzed (Participants) | 96 | 104
percentage of participants | 73.7 | 83.1

2. Secondary Outcome: The Percentage of Participants With Retention Rate
Description: The percentage of participants who completed the trial.
Time Frame: 24 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Zonisamide | Carbamazepine
Number analyzed (Participants) | 96 | 104
percentage of participants | 59.4 | 62.5

3. Secondary Outcome: Quality of Life in Epilepsy (QoL-QOLIE31)
Description: Quality of life assessment tool. Overall scores is calculated by summing subsections, and it ranges from 0 to 100. Higher score presents higher quality of life.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: Units On a Scale
Arm/Group | Zonisamide | Carbamazepine
Number analyzed (Participants) | 96 | 104
Units On a Scale
  Pre-QOLIE 31 | 60.72 (14.69) | 61.96 (16.67)
  Post-QOLIE 31 | 67.27 (16.34) | 69.51 (17.61)

ADVERSE EVENTS:
Arm/Group | Zonisamide | Carbamazepine
Serious Adverse Events (participants affected / at risk) | 5/96 | 9/104
Other Adverse Events (participants affected / at risk) | 74/96 | 70/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zonisamide (N=96) | Carbamazepine (N=104)
Worsening Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Depressive Mood (Psychiatric disorders) | 1 (1) | 0 (0)
Right Shoulder Injury (General disorders) | 1 (1) | 0 (0)
Visual Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Cervical Sprain (General disorders) | 1 (1) | 0 (0)
Memory And Judgement Disturbance (Psychiatric disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Uterine Fibroid (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Sgpt Increased (Investigations) | 0 (0) | 1 (1)
Sgot Increased (Investigations) | 0 (0) | 1 (1)
Mental Torpor (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zonisamide (N=96) | Carbamazepine (N=104)
Dizziness (Nervous system disorders) | 28 (30) | 23 (24)
Drowsiness (Psychiatric disorders) | 25 (25) | 24 (25)
Anorexia (Gastrointestinal disorders) | 20 (21) | 5 (5)
Weight Decrease (Investigations) | 16 (17) | 2 (2)
Headache (Nervous system disorders) | 14 (14) | 14 (14)
Nausea (Gastrointestinal disorders) | 11 (11) | 12 (14)
Memory Impairment (Psychiatric disorders) | 9 (9) | 5 (5)
Mental Torpor (Psychiatric disorders) | 7 (7) | 12 (12)
Gastrointestinal Pain (Gastrointestinal disorders) | 7 (7) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (7) | 4 (5)
Sleep Disorder (Psychiatric disorders) | 6 (6) | 4 (4)
Fatigue (General disorders) | 7 (7) | 6 (6)
Pyrexia (General disorders) | 6 (6) | 8 (9)
Rash (Skin and subcutaneous tissue disorders) | 6 (6) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 5 (6) | 2 (2)
Depression (Psychiatric disorders) | 4 (4) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5)
Constipation (Gastrointestinal disorders) | 1 (1) | 7 (7)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 6 (7)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No